CLINICAL TRIAL: NCT06198673
Title: Real-world Patterns of Anti-platelet Management in Stable Angina Patients Undergoing Percutaneous Coronary Intervention
Brief Title: A Prospective muLticEnter Registry in chrONic coronARy synDrOme
Acronym: LEONARDO
Status: Not yet recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, PROFESSOR OF CARDIOLOGY, University of Roma La Sapienza
Other Study IDs: 2023/D/18122023
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Platelet Aggregation Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antiplatelet Agents — Antiplatelet agents more commonly used at time of percutaneous coronary intervention in patients with chronic coronary syndrome

SUMMARY:
In patients with chronic coronary syndrome (CCS), clopidogrel has a class I/A indication in patients undergoing elective percutaneous coronary intervention (PCI). Although unproven, the possibility exists that clopidogrel does not yield an optimal platelet inhibition in multiple real-world scenarios that challenge current recommendations.

The aim of this prospective observational study io assess in a consecutive unselected series of patients with CCS undergoing elective PCI the frequency of the following real world clinical scenarios:

* No pretreatment at time of PCI ('naïve')
* Evidence of incomplete responsiveness to clopidogrel
* Indication to a complex PCI.

We expect to demonstrate:

* A not negligible proportion of patients with CCS are 'naïve' at time of elective PCI in clinical practice and require a rapid onset of P2Y12 inhibition.
* A substantial proportion of patients with CCS who are treated with clopidogrel prior to elective PCI have high platelet responsiveness at time of the procedure.
* A complex PCI is performed in a substantial proportion of patients with CCS.

DETAILED DESCRIPTION:
In patients with chronic coronary syndrome (CCS), clopidogrel has a class I/A indication in patients undergoing elective percutaneous coronary intervention (PCI) (Figure 1). Initiation of oral P2Y12 inhibitors is usually delayed until the coronary anatomy is defined (Knuuti, Levine). Clopidogrel (administered as a 600 mg loading dose followed by a 75 mg maintenance dose) is the P2Y12 inhibitor of choice in CCS patients undergoing PCI (Knuuti, Levine). Also, pre-treatment with clopidogrel is currently recommended if the probability of PCI is high (II B/C). Although unproven, the possibility exists that clopidogrel does not yield an optimal platelet inhibition in multiple real-world scenarios that challenge current recommendations, as follows:

* P2Y12 inhibitors 'naive' patients with CCS who have an indication to PCI after coronary angiography might experience deferral of PCI because they are not pre-treated with clopidogrel (Selvarajah, 2021)
* Heterogeneity in individual response profiles to clopidogrel, with a considerable number of patients yielding inadequate platelet inhibitory effects, might result in increased risk of thrombotic events post-PCI (Galli). Individual responsiveness to P2Y12 inhibitors can be assessed through platelet function testing (Franchi), but its implementation in clinical practice is currently not recommended. As a consequence, a significant proportion of CCS patients are not on a fully effective dual antiplatelet therapy (DAPT) at time of PCI.
* Complex PCIs are increasingly performed in CCS patients. Complex PCI is commonly defined by any of the following characteristics: ≥ 3 drug eluting stents implanted, bifurcation PCI with 2 stents, left main coronary artery PCI, saphenous vein graft PCI, total stent length > 60 mm, or chronic total occlusion as target lesion (Figure 2). Importantly, patients who undergo complex PCI have a substantially higher ischemic risk with increased procedural complexity (Giustino, Genereaux). Preliminary observations suggest that an intensive periprocedural platelet inhibition, even on top of DAPT pretreatment, might be of benefit in stable patients undergoing percutaneous revascularization of complex lesions (Marchese).

To assess in a consecutive unselected series of patients with CCS undergoing elective PCI the frequency of the following real world clinical scenarios:

* No pretreatment at time of PCI ('naïve')
* Evidence of incomplete responsiveness to clopidogrel
* Indication to a complex PCI Consecutive patients with CCS undergoing elective PCI.

Patients will be grouped as follows:

* Pre-treatment with clopidogrel before elective PCI
* Patients receiving a clopidogrel loading at time of elective PCI in the cath lab Patients receiving cangrelor during PCI in the cath lab and then receiving a P2Y12 inhibitor afterwards
* Patients with CCS undergoing elective PCI
* Patients' written informed and privacy consent obtained before the PCI procedure
* Male or female patients 18 to 80 years old
* Assessment of response to anti-platelet agents by VerifyNowTM
* Patients with active bleeding
* Patients with hypersensitivity to any anti-platelet agents or to any of its excipients
* Known pregnancy or breast-feeding female patients > 1,000 patients Multicenter evaluation
* Pre-treatment with clopidogrel before elective PCI
* Patients receiving a clopidogrel loading at time of elective PCI in the cath lab
* Patients receiving cangrelor during PCI in the cath lab and then receiving a P2Y12 inhibitor afterwards

  1-year
  1. Frequency of 'naive' patients with CCS undergoing elective PCI
  2. Frequency of complex coronary intervention in patients undergoing elective PCI
* Frequency of incomplete response to clopidogrel prior to elective PCI (as assessed by VerifyNow TM)
* Frequency of the use of periprocedural i.v. cangrelor
* Frequency of the use of glycoprotein IIb/IIIa (GPIIb/IIIa) inhibitors
* Frequency of the use of clopidogrel, ticagrelor or prasugrel loading dose
* Mode of administration of oral P2Y12 inhibitors (crushed)
* Incidence of post-PCI ischemic complications
* Incidence of any post-PCI bleeding according to the Bleeding Academic Research Consortium [BARC] criteria
* Incidence of major adverse cardiac events (MACE) - MACE will comprise any of the following events: death, myocardial infarction (MI), ischemia-driven revascularisation (IDR) and stent thrombosis (ST)
* Enrolment phase (1 year)
* Follow-up: 1-year

The study will be conducted in accordance with the Declaration of Helsinki on ethical principles for medical research involving human subjects.

Informed consent to be included in this survey is mandatory for collecting individual data and must be obtained from all subjects and/or their legal representative(s) as per local regulations.

We expect to demonstrate:

* A not negligible proportion of patients with CCS are 'naïve' at time of elective PCI in clinical practice and require a rapid onset of P2Y12 inhibition.
* A substantial proportion of patients with CCS who are treated with clopidogrel prior to elective PCI have high platelet responsiveness at time of the procedure.
* A complex PCI is performed in a substantial proportion of patients with CCS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CCS undergoing elective PCI
* Patients' written informed and privacy consent obtained before the PCI procedure
* Male or female patients 18 to 80 years old
* Assessment of response to anti-platelet agents by VerifyNowTM

Exclusion Criteria:

* Patients with active bleeding
* Patients with hypersensitivity to any anti-platelet agents or to any of its excipients
* Known pregnancy or breast-feeding female patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with CCS undergoing elective PCI.
  Patients will be grouped as follows:
  * Pre-treatment with clopidogrel before elective PCI
  * Patients receiving a clopidogrel loading at time of elective PCI in the cath lab Patients receiving cangrelor during PCI in the cath lab and then receiving a P2Y12 inhibitor afterwards
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of 'naive' patients with CCS undergoing elective PCI | up to 12 months
  Number of 'naive' patients with CCS undergoing elective PCI
Frequency of complex coronary intervention in patients undergoing elective PCI | up to 12 months
  Number of complex coronary intervention in patients undergoing elective PCI

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pelliccia, MD, Principal Investigator — University Sapienza

IPD SHARING:
Plan to Share IPD: Undecided